CLINICAL TRIAL: NCT05126160
Title: Immune Score Based Radiomics in Nasopharyngeal Carcinoma (IMRAN Study)
Brief Title: Immune Score Based Radiomics in Nasopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZJCH-2021-NPC01
Record Dates: First submitted 2021-11-07; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immune Score Based Radiomics — To establish an immune score based radiomic staging system for nasopharyngeal carcinoma

SUMMARY:
In nasopharyngeal carcinoma (NPC), tumor, node and metastasis (TNM) staging system is the main tool for determining treatment strategy and assessment of prognosis. However, the prognoses of patients with the same TNM stage after similar treatment vary widely. The aim of this study is to establish an immune score based radiomic staging system for NPC.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly histologically confirmed non-keratinizing/keratinizing carcinoma.

ECOG Performance status: 0-1 With normal liver function test (ALT, AST ≤2.5ULN) Renal: creatinine clearance ≥60ml/min Without hematopathy,marrow: WBC >4*109/L, HGB>90G/L, and PLT>100*109/L. Written informed consent

Exclusion Criteria:

Contraindications for MRI scan Prior malignancy (except adequately treated carcinoma in-situ of the cervix or · basal/squamous cell carcinoma of the skin) Previous chemotherapy or radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume) Patient is pregnant or lactating Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), or emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-metastatic NPC patients receive radical radiotherapy with/without induction or concurrent chemotherapy. De novo metastatic NPC patients would receive at least 4 cycles of platinum-based therapy.
Sampling Method: Probability Sample
Enrollment: 494 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Median follow-up time of 5 years for the whole group
  The AUC of the immune score based radiomic staging system

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, Principal Investigator — Department of Radiation Oncology, Zhejiang Cancer Hospital
Locations (5):
- China (5):
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Ningbo First Hospital, Ningbo, Ningbo
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Ningbo
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Wenzhou
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided